CLINICAL TRIAL: NCT04733807
Title: Sars-Cov2 Antibodies Response to vaccinE Against covId-19 Disease
Brief Title: Antibodies Response to mRNA Vaccine Against Covid-19
Acronym: SCAREAID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: ICOT University Hospital (Unknown)
Responsible Party: Principal Investigator, Luigi Iuliano, Professor of Internal Medicine, University of Roma La Sapienza
Other Study IDs: SCAREAID
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Covid-19
Keywords: vaccine; Covid-19; safety; Sars-Cov2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: BNT162b2 mRNA Covid-19 Vaccine — Hospital employers vaccinated with BNT162b2 mRNA against Sars-Cov2 are studied for serum antibody response.

SUMMARY:
Vaccine rollout has started in many countries. In Italy, the Covid-19 vaccine used at the moment is the mRNA-based BNT162b2 and is given to Hospital employers. The investigators undertake this study to monitor IgG evolution after vaccination in the participant hospital settings, which includes 500 subjects.

DETAILED DESCRIPTION:
Vaccine rollout has started in many countries. In Italy, the Covid-19 vaccine used at the moment is the mRNA-based BNT162b2 and is given to Hospital employers.

The investigators undertake this observational study to monitor antibody evolution after vaccination in a hospital setting. The primary endpoint is serum IgG at the first month of 2nd jab, and at 3, 6, and 12 months afterward.

As secondary measures, nasopharyngeal swabs are included, at fortnight intervals to detects the spike protein antigen, in the event that putative vaccine inefficacy would expose the health personnel to Covid-19 disease with potential spreading to inpatients.

Further, clinical signs and symptoms are monitored at the weekly interval in the context of adverse reactions/events.

ELIGIBILITY:
Inclusion Criteria:

* Hospital employers vaccinated against Sars-Cov2

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health care, administrative, and technical workers of ICOT-Sapienza University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Serum IgG antibodies levels in response to vaccine | Serum antibody at 1 month
  Determination of IgG levels in serum
Serum IgG antibodies levels in response to vaccine | Serum antibody at 3 months
  Determination of IgG levels in serum
Serum IgG antibodies levels in response to vaccine | Serum antibody at 6 months
  Determination of IgG levels in serum
Serum IgG antibodies levels in response to vaccine | Serum antibody at 12 months
  Determination of IgG levels in serum

SECONDARY OUTCOMES:
Sars-Cov2 infection in vaccinated subjects | up to 12 months
  Monitoring of Sars-Cov2 infection by a nasopharyngeal swab of spike protein Ag, and PCR confirmation in case of Ag swab positivity.
Covid-19 disease in vaccinated subjects | Clinical monitoring of vaccinated subjects through the study completion, an average of 1 year.
  Monitoring the occurrence of Covid-19 disease in vaccinated people

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Iuliano, M.D., Principal Investigator — University of Roma La Sapienza
Locations (1):
- ICOT-Sapienza University Hospital, Latina, LT, Italy

IPD SHARING:
Plan to Share IPD: Undecided